CLINICAL TRIAL: NCT05721092
Title: Assessment of Knowledge, Facilitators and Barriers of Pneumococcal Vaccination: A Cross-sectional Study Among Diabetologists in India
Brief Title: Assessment of Knowledge on Pneumococcal Vaccination Among Diabetologists in India
Status: Completed | Type: Observational
Sponsor: M.V. Hospital for Diabetes (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, Vijay Viswanathan, Managing Director, M.V. Hospital for Diabetes
Other Study IDs: 2023_01_MSDMVH
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Pneumococcal Vaccine
MeSH Terms: interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pre and Post Education on practice of pneumococcal vaccination — A cross-sectional study will be conducted among 25 diabetologists in each of the four zones in India representing all directions - North, East, West and South. Diabetologists will be selected through purposive sampling. A semi-structured questionnaire (study tool) is designed based on the existing literature that addresses our objectives. An education session on Pneumococcal vaccination will be conducted for the diabetologists through webinar after completing the survey. A post assessment will be done using the same questionnaire among the study participants after the education session in order to see an increase in the knowledge of pneumococcal vaccination.

SUMMARY:
Asia has the highest burden with the largest contribution of pneumonia burden from India. Pneumonia is also observed as 5th leading cause of deaths in India. People with diabetes with uncontrolled glucose are significantly at higher risk of development of pneumonia. Even though, pneumonia is a vaccine-preventable disease, hospitalization for pneumonia of patients with diabetes are rising. Very limited literature is available on the knowledge and practice of pneumonia vaccination among diabetologists and the rate of pneumonia vaccination received by the patients with diabetes. Hence this study aims to assess their knowledge on the same. In addition, this study also aims to identify the real barriers and facilitators of pneumococcal vaccination among diabetologists in India. A cross-sectional study will be conducted among 25diabetologists in each of the four zones in India representing all directions - North, East, West and South. Diabetologists will be selected through purposive sampling. A semi-structured questionnaire (study tool) is designed based on the existing literature that addresses our objectives. An education session on Pneumococcal vaccination will be conducted for the diabetologists through webinar after completing the survey. A post assessment will be done using the same questionnaire among the study participants after the education session in order to see an increase in the knowledge of pneumococcal vaccination.

ELIGIBILITY:
Inclusion Criteria:

Diabetologists willing to participate in the study

Exclusion Criteria:

Unwillingness to give consent for participation

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetologists aged 25 to 65, practicing in India
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
To identify the facilitators and barriers of pneumococcal vaccination among diabetologists in India. | 6 months

SECONDARY OUTCOMES:
To assess the knowledge, attitude and practices of pneumococcal vaccination among select diabetologists across India. | 6 months
To examine the association of knowledge and practice of vaccination among diabetologists | 6 months
To assess the change in the knowledge of pneumococcal vaccination post educational intervention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Viswanathan, Principal Investigator — M V Hospital for Diabetes [P] Limited
Locations (1):
- M V Hospital for Diabetes [P] Limited, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No